CLINICAL TRIAL: NCT03571035
Title: Presentation of Light and Affordable Vision System for Mandibular Trajectory Assessment in Women With Mild Temporomandibular Joint Disorder
Brief Title: The Vision System for Mandibular Trajectory Assessment in Women With Mild Temporomandibular Joint Disorder
Acronym: UMP14/06
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jagoda Goślińska, Principal Investigator, Poznan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 501/14
Record Dates: First submitted 2018-06-17; First posted 2018-06-27 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Mandibular Deviation
Keywords: Mandibular deviation; mandibular movement recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Example (Experimental): Mandibular movements recordings by a mono vision system.
  Interventions: Diagnostic Test: Mandibular movements recordings by a mono vision system

INTERVENTIONS:
Diagnostic Test: Mandibular movements recordings by a mono vision system — To examine the mandible's movements, vision analysis was employed and performed with the digital camera which featured 1920 x 1080 resolution and was fixed on an aluminium extension arm attached to a headset worn by the subject.The camera was aligned parallel to the subject's face at a distance of 0.3 meters. The study used two 10 mm x 5 mm reference markers, which were accurately reproduced on the camera recorded images. In line, one marker was put on the medial cleft above the upper lip, and the other one was positioned below the first one in a straight line, in the middle of the chin. Then, the patient was asked to open maximally and close the mouth twice.To establish the mandible's trajectory, the line was drawn between the positions of the two markers to connect the two points. The line's parameters were calculated only during initial measurements and were constant throughout the study.

SUMMARY:
Recording mandibular movements plays an important role in stomatognathic system diagnosis and has been the subject of numerous research projects. This study presents theoretical assumptions and a practical solution in the form of a novel method of mandibular motion assessment.

DETAILED DESCRIPTION:
In the presented method, mandibular movements are recorded by a mono vision system where a digital camera is fixed on a special extension arm attached to patient's head. During movement the camera records changing positions of two markers placed on two selected two points on a patient's face. With such data, it possible to assess the absolute range of mandibular abduction as well as displacements from optimal trajectory occurring during movement, which indicative of stomatognathic dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* temporomandibular joint disorder
* qualitative and quantitative impairments of mandibular movements

Exclusion Criteria:

* no impairments of mandibular movements

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
Range of mandibular abduction [mm] | about 2 minutes
  The maximum mouth opening value calculated as the difference in the distance between the markers before registration and during the maximum opening.
Maximum displacement in frontal plane [mm] | about 2 minutes
  The value of the maximum deviation of the lower marker in relation to the upper one in the frontal plane.
Normalized displacement in frontal plane [mm^2/s] | about 2 minutes
  The value of normalized displacement calculated by dividing the sum of squared errors in movement trajectory on the transverse axis by the number of measurements taken during analysis time.

CONTACTS AND LOCATIONS:
Overall Officials: Przemysław Lisiński, PhD, Study Director — Poznań University of Medical Sciences